CLINICAL TRIAL: NCT01344720
Title: Evaluation of the Efficacy and Tolerability of Etoricoxib Monotherapy Versus Combination Oxycodone-etoricoxib in Moderate to Severe Pain From Chronic Low Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria Locale 4, Teramo (Other)
Responsible Party: Dott. Pier Luigi Orsini, Dipartimento Emergenza ed Accettazione Ospedale Civile G. Mazzini Teramo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASL 4 Teramo
Record Dates: First submitted 2011-04-13; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-03

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Etoricoxib; Oxycodone
MeSH Terms: conditions — Low Back Pain | interventions — Etoricoxib; Oxycodone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- etoricoxib (Active Comparator): etoricoxib up to 60mg/day as monotherapy
  Interventions: Drug: etoricoxib
- etoricoxib plus controlled-release oxycodone (Active Comparator): combination treatment of etoricoxib (30 mg/day) plus controlled-release oxycodone (10 mg/day)
  Interventions: Drug: oxycodone

INTERVENTIONS:
Drug: etoricoxib — At visit 2 eligible patients will then receive Etoricoxib 30mg for 2 weeks. Patients who achieve a clinically meaningful improvement in pain at the end of this period (defined as a ≥30% improvement in BPI avg daily pain intensity), will continue therapy up to week 5 (visit 4), if they become "non-responders" between week 4-5, they can be tapered off meds and then discontinued from the study. Patients who do not achieve a clinically meaningful improvement will be considered "non-responders" and will be randomized to receive either titration of their monotherapy or combination treatment.
  Group 1 "non-responders" will receive an increase in monotherapy from etoricoxib 30mg to eterocoxib 60mg/die.
  Arms: etoricoxib
Drug: oxycodone — At visit 2 eligible patients will then receive Etoricoxib 30mg for 2 weeks. Patients who achieve a clinically meaningful improvement in pain at the end of this period (defined as a ≥30% improvement in BPI avg daily pain intensity), will continue therapy up to week 5 (visit 4), if they become "non-responders" between week 4-5, they can be tapered off meds and then discontinued from the study. Patients who do not achieve a clinically meaningful improvement will be considered "non-responders" and will be randomized to receive either titration of their monotherapy or combination treatment.
  Group 2 "non-responders" will receive in addition to etoricoxib 30mg/day a dose of oxycodone CR 5mg q12hr (dose of 5mg tablet is available in Italy).
  Arms: etoricoxib plus controlled-release oxycodone

SUMMARY:
This randomized, single-blind, parallel-group study will investigate the efficacy and the tolerability of a combination treatment of etoricoxib (30 mg/day) plus controlled-release oxycodone (10 mg/day) compared with a titrated dose of etoricoxib up to 60mg/day as monotherapy , in patients with Chronic Low Back Pain (CLBP) who have not responded to the starting dose of Etoricoxib 30mg/day. A common clinical question is that is it better to increase the dose of the current monotherapy or to combine both treatments early on, in patients who do not respond to standard start doses of NSAIDs like etoricoxib.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients (at least 18 years of age).
* Patient with a confirmed diagnosis of moderate-to-severe CLBP present for more than 15 days per month and several hours per day for at least 6 months prior to screening.
* Achieve at least 3 consecutive days with an average daily pain score > 4 during baseline week (between visit 1 and visit 2) via patient diary recordings.
* Patient is currently not receiving treatment for CLBP or was receiving treatment for CLBP, with a drug other than etoricoxib or oxycodone, and completed the required washout prior to Visit 2.
* Patient has never received treatment with etoricoxib or oxycodone and other strong opioids.
* No assumption of adjuvant drugs (antiepileptics, steroids, tricyclic antidepressants, SNRIs, muscle relaxants) in the last month (or two week).
* Patient has a level of understanding sufficient to provide written informed consent and to communicate with the investigator and site personnel.
* Patient is judged to be reliable, agrees to keep all appointments for clinic visits, and agrees to participate in recording responses to questionnaires and other instruments used in this study, as well as all other protocol procedures.
* All females of child-bearing potential must test negative for pregnancy at Visit 1, based on a serum pregnancy test. Females of child-bearing potential (not surgically sterilised and between menarche and 1 year post-menopause) must agree to use a medically acceptable and reliable means of birth control (as determined by the investigator) during the study and for 1 month following the last dose of study drug. Examples of reliable methods include use of oral contraceptives or Depo Provera Contraceptive Injection, abstinence, partner with vasectomy, diaphragm with contraceptive jelly, condom with contraceptive foam, and intrauterine devices.

Exclusion Criteria:

* Have a known hypersensitivity to NSAIDs or strong opioids or any of the inactive ingredients or have any contraindication for the use of etoricoxib or oxycodone:
* Patient with hypersensitivity to opioid analgesics;
* acute asthma or other obstructive airway disease and acute respiratory depression with hypoxia;
* elevated carbon dioxide levels in the blood; cor pulmonale; acute alcoholism; delirium tremens;severe CNS depression; convulsive disorders; increased cerebrospinal or intracranial pressure;
* head injury; suspected surgical abdomen (paralytic ileus); concomitant MAO inhibitors (or within 14 days of such therapy).
* Hypersensitivity to the active substance or to any of the excipients of etoricoxib formulation.
* Active peptic ulceration or active gastro-intestinal (GI) bleeding.
* Patients who have experienced bronchospasm, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria, or allergic-type reactions after taking acetylsalicylic acid or NSAIDs including COX-2 (cyclooxygenase-2) inhibitors.
* Pregnancy and lactation
* Severe hepatic dysfunction (serum albumin <25 g/l or Child-Pugh score ≥10).
* Estimated renal creatinine clearance <30 ml/min.
* Inflammatory bowel disease.
* Congestive heart failure (NYHA II-IV).
* Patients with hypertension whose blood pressure is persistently elevated above 140/90mmHg and has not been adequately controlled.
* Established ischaemic heart disease, peripheral arterial disease, and/or cerebrovascular disease.
* Have previously completed or withdrawn from this study or any other study investigating etoricoxib or oxycodone or have previously been treated with etoricoxib or oxycodone.
* Have a history of substance abuse or dependence within the past year, excluding nicotine and caffeine.
* Have a positive urine drug screen for substances of abuse. Women who are breast-feeding.
* Have a historical exposure to drugs known to cause neuropathy (for example, vincristine), or a history of a medical condition, including pernicious anaemia and hypothyroidism, that could have been responsible for neuropathy.
* Have pain that cannot be clearly differentiated from or conditions that interfere with the assessment of the CLBP. Examples of painful conditions that could be confused like peripheral vascular disease (ischemic pain); neurological disorders (for example, phantom limb pain from amputation); skin condition in the area of the neuropathy that could alter sensation (for example, plantar ulcer); other painful conditions (for example, arthritis, neoplasm, fibromyalgia, CRPS).
* Have a history of neurosurgical procedures for pain control, nerve/plexus blocs or ablation within 6 months prior to screening.
* Psychological conditions that, in the opinion of the investigator, would compromise participation or be likely to require hospitalization during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a > 30% reduction in avg daily pain intensity at treatment week 4 (Visit 4). | from baseline (avg of daily diary scores between visit 1 and 2) to the end of treatment week 5
  Proportion of patients achieving a > 30% reduction in avg daily pain intensity at treatment week 4 (Visit 4). Pain will be measured by the mean change of question #5 (avg daily pain intensity) of the Brief Pain Inventory (BPI) Modified Short Form from baseline (avg of daily diary scores between visit 1 and 2) to the end of treatment week 5 (Visit 4).

SECONDARY OUTCOMES:
Proportion of patients achieving a > 50% reduction in avg daily pain intensity at treatment week 5 (visit 4). | from baseline (avg of 3 qualifying days from diary scores between visit 1 and 2) to the end of treatment week 5
  1. Proportion of patients achieving a > 50% reduction in avg daily pain intensity at treatment week 5.
  2. Proportion of patients achieving a > 30% reduction in avg daily pain intensity at treatment week 3 (visit 3).
  3. Average daily change in pain intensity from baseline to treatment week 5
  4. Average daily change in pain intensity from baseline to treatment week 3
  5. Mean change in CLBP Disability from baseline to end of treatment week 5

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Orsini, Dottore, Principal Investigator — Dipartimento Emergenza ed Accettazione Ospedale Civile G. Mazzini Teramo
Locations (5):
- Italy (5):
  - Dipartimento di Scienze della Salute Anestesia, Rianimazione e Terapia del dolore - Università degli Studi di L'Aquila Ospedale San Salvatore L'Aquila, L’Aquila, L'Aquila
  - Unità di riabilitazione neurofisiologica Istituto Scientifico di Riabilitazione di Montescano, Montescano (PV), Pavia
  - Clinica Anestesia e Rianimazione Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma, Roma
  - Dipartimento Emergenza ed Accettazione Ospedale Civile G. Mazzini Teramo, Teramo, Teramo
  - Dipartimento di Medicina Interna- Università degli Studi di Perugia Azienda Ospedaliera S.Maria - Clinica Medica, Terni, Terni